CLINICAL TRIAL: NCT05809713
Title: Carolina Consortium for Improved BP Control in Vulnerable Populations
Brief Title: Heart to Heart: BP Control Partners
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IHS-2021C3-25060
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology enabled Team Care (Experimental): Ongoing Team-based, Pharmacist led telephonic management of uncontrolled high blood pressure involving cellular-enabled home BP monitoring, medications, diet and exercise, and referral for social problems
  Interventions: Other: Technology-enabled Team Care
- Enhanced Usual Care (Active Comparator): Home BP monitoring device provided along with BP log, basic diet and exercise instruction, and care provided by the patient's usual doctor/provider
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Other: Technology-enabled Team Care — Patients randomized to the TTC arm will receive telehealth-enabled team-based care. The team will include a physician and/or advanced practice provider, a pharmacist with Certified Pharmacist Practitioner (CPP) status or similar skills in NC, and will incorporate brief nutritionist-directed lifestyle behaviors counseling (DASH diet; exercise) initially delivered every other week by phone for two months, followed by monthly calls (once SBP values achieve individualized goal and remain stable for 14 days) over 12 months supported by cellular enabled home BP monitoring.
  Arms: Technology enabled Team Care
Other: Enhanced Usual Care — Patients randomized to the enhanced usual care (EUC) arm will receive telehealth enabled home BP monitoring equipment including set-up and instruction and basic hypertension-specific lifestyle (diet, exercise) instruction and materials at baseline, but will not receive telehealth-enabled team-based care, active home BP monitoring by a pharmacist, or detailed DASH intensive lifestyle counseling.
  Arms: Enhanced Usual Care

SUMMARY:
The goal of this clinical trial is to compare a new model of care that uses cellular-enabled home blood pressure (BP) telemonitoring and combines it with team-based BP control using a pharmacist to help manage BP medications and to give patients advice on diet and exercise, to an enhanced usual care group that only receives the monitoring device and basic instructions, in individuals with a history of uncontrolled hypertension. The main question[s] it aims to answer are:

1. Among patients with a history of uncontrolled hypertension, evaluate the impact of team-based care using technology-enabled monitoring on improving goal-directed systolic blood pressure (SBP) levels relative to enhanced usual care (primary).
2. Assess the potential for heterogeneity of treatment effects by race, age, sex, and social deprivation index (secondary).
3. Examine the impact of the intervention on hypertension self-efficacy, medication adherence, timeliness of medication change, satisfaction with care, adoption of home BP monitoring, and the change in mean BP in diverse patients, many of whom have adverse social determinants of health (SDOH) (secondary/exploratory).

Both groups will be asked to check their BP at home using a cellular-enabled home BP monitoring device that's provided. Patients in the Technology enabled Team Care (TTC) intervention group will have regular phone calls from a clinically trained and experienced pharmacist that works with their doctor/provider and who has reviewed their home BP readings. This pharmacist will help them adjust their medicines, provide brief nutrition and physical activity advice, and may refer them for help with any social challenges (not enough proper food, transportation problems, etc.) that they may be experiencing. An enhanced usual care group will serve as the comparison group and will receive the BP cuff monitoring device and basic instructions but will not receive ongoing monitoring or team care as described above.

Researchers will compare the effect of the TTC intervention model to enhanced usual care to assess the impact on SBP levels at 6 and 12 months follow-up, as well as on a variety of patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic and non-Hispanic black (≥50%) and white (≤50%) adults (>18yr. old; 40% male)
* diagnosis of essential hypertension,
* a documented history of uncontrolled hypertension (mean SBP ≥ 140 mmHg from primary care office visits over the last year) and
* elevated SBP (≥ 140 mmHg) (average of 2 research-grade measurements) at the time of enrollment.

Exclusion Criteria: Patients with:

* severe chronic kidney disease (eGFR < 30 ml/min/1.73m2),
* substance abuse,
* difficulty with communication in English without an interpreter,
* dementia, mental illness or any condition that would limit ability to give informed consent
* rare patients living in very remote areas where cellular- enabled telemonitoring is not feasible will be excluded.
* Pregnancy; female participants will be asked to report pregnancy status during pre-screening and at study baseline. Participants who report pregnancy prior to randomization will be excluded from the study. If the participant becomes pregnant during the study, prescribed medication(s) will be rapidly tapered or immediately discontinued, as indicated and the patient referred back to their primary care provider for follow-up.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure (SBP) level at 6 months follow-up | 6-months
  Change from baseline visit to six-months follow-up visit in measured SBP

SECONDARY OUTCOMES:
Change in Systolic Blood Pressure (SBP) level at 12 months follow-up | 12 months
  Change from baseline visit to 12-months follow-up visit in measured SBP
Improved SBP Control at 6 and 12 months | 6 and 12 months follow-up
  Proportion with SBP < 140 mmHg in TTC intervention vs. enhanced usual care (EUC) pts. at 6 and 12 mo.

CONTACTS AND LOCATIONS:
Overall Officials: Doyle Cummings, Pharm.D., Principal Investigator — East Carolina University Brody School of Medicine
Locations (2):
- United States (2):
  - ECU Family Medicine Center, Greenville, North Carolina
  - Cape Fear Clinic, Wilmington, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided
Investigators will work with IRB and study sponsors to define a data sharing plan